CLINICAL TRIAL: NCT04775082
Title: Effect and Safety of Liraglutide 3.0 mg on Weight Management in Children With Obesity Aged 6 to Below 12 Years: 56-week, Double-blind, Randomised, Placebo-controlled Trial
Brief Title: SCALE KIDS: Research Study to Look at How Well a New Medicine is at Lowering Weight in Children With Obesity
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN8022-4392; U1111-1247-8226 (Other: World Health Organization (WHO)); 2020-000546-34 (Registry Identifier: European Medicines Agency (EudraCT))
Record Dates: First submitted 2021-02-26; First posted 2021-03-01 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Liraglutide 3.0 mg (Experimental): The treatment duration is 56 weeks and the follow-up period is 26 weeks.
  Interventions: Drug: Liraglutide
- Placebo (Placebo Comparator): The treatment duration is 56 weeks and the follow-up period is 26 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Liraglutide — The study medicine must be injected in a skin fold in the stomach, thigh or upper arm once daily.
  The dose will increase each week over 4 or 5 weeks until the final dose is reached.
  Arms: Liraglutide 3.0 mg
Drug: Placebo — The study medicine must be injected in a skin fold in the stomach, thigh or upper arm once daily.
  Arms: Placebo

SUMMARY:
The study looks at how liraglutide works on participant's body weight. Researchers will look at how liraglutide can help children with obesity to lose weight. They will look at how much weight the children will lose, and if there are any side effects.

Participants will either get liraglutide or placebo. Which treatment the participants get is decided by chance. Liraglutide is a new medicine for children, but it can already be prescribed by doctors to adults with overweight or obesity. The participant will get 1 injection every day.

In addition to taking the medicine, the participants will have talks with the study staff about healthy food choices, how they can be more physically active and what can be done to help the participants to lose weight.

The study will last for about 96 weeks (almost 2 years). The participants will have 18 clinic visits and 10 phone or video calls with the study doctor/staff. Participant will have blood samples taken, have 1 test to check the heart, 1 hand X-ray taken and must fill in a diary between some of the visits.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent of parent(s) or legally acceptable representative of subject and child assent, as age-appropriate, obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial
* Male or female, aged 6 to below 12 years at the time of signing informed consent
* Tanner stage 1-5 pubertal development at the time of signing informed consent
* BMI above or equal to 95th percentile, on gender and age-specific growth charts (CDC.gov)
* History of failing to lose sufficient weight with lifestyle modification as judged by the investigator

For subjects with type 2 diabetes at screening the following inclusion criterion apply in addition:

- Hemoglobin A1c (HbA1c) below or equal to 10.0 percent (86 mmol/mol) as measured by central laboratory at screening

Exclusion Criteria:

* A self-reported (or by parent(s)/LAR (legally acceptable representative) where applicable) change in body weight above 5 kg (11 lbs) within 90 days before screening irrespective of medical records
* Treatment with any medication for the indication of obesity within the past 90 days before screening
* Type 1 diabetes
* Subjects with secondary causes of obesity (for example hypothalamic, monogenic or endocrine causes)

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Estimated)
Dates: Start 2021-03-04 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Relative change in BMI (Body mass index) | From baseline (week 0) to week 56
  Percent

SECONDARY OUTCOMES:
Relative change in body weight | From baseline (week 0) to week 56
  Percent
Change in BMI standard deviation score (WHO.int) | From baseline (week 0) to week 56
  Unitless
Subjects achieving above or equal to 5 percent reduction of BMI | From baseline (week 0) to week 56
  Yes/no
Subjects achieving above or equal to 10 percent reduction of BMI | From baseline (week 0) to week 56
  Yes/no
BMI percentage of the 95th percentile on gender and age-specific growth charts (CDC.gov) | From baseline (week 0) to week 56
  Percent point
Change in waist circumference | From baseline (week 0) to week 56
  cm
Change in systolic blood pressure | From baseline (week 0) to week 56
  mmHg
Change in diastolic blood pressure | From baseline (week 0) to week 56
  mmHg
Change in HbA1c (glycated haemoglobin) | From baseline (week 0) to week 56
  Percent point
Treatment emergent adverse events (TEAEs) | From baseline (week 0) to week 82
  Number
Treatment emergent serious adverse events (SAEs | From baseline (week 0) to week 82
  Number

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (31):
- United States (9):
  - TMC Hlthcr Clin Res Office, Tucson, Arizona
  - Children's Hospital Colorado, Denver, Colorado
  - Solaris Clinical Research, Meridian, Idaho
  - Pennington Biom Res Ctr, Baton Rouge, Louisiana
  - Barry J. Reiner, MD LLC, Baltimore, Maryland
  - University of Minnesota_CPOM, Minneapolis, Minnesota
  - UBMD Peds-Div of Endo/Diabetes, Buffalo, New York
  - PriMed Clinical Research, Dayton, Ohio
  - UPMC Child Hosp-Pittsburgh, Pittsburgh, Pennsylvania
- Belgium (2):
  - UZ Brussel, Brussels
  - UZ Leuven - Kindergeneeskunde, Leuven
- India (2):
  - Endolife Specialty Hospitals, Guntur, Andhra Pradesh
  - Mamc & Lnjp, New Delhi
- Israel (2):
  - Rambam MC - Department of Pediatrics A, Haifa
  - Schneider MC - Endrocrinology and Diabetes, Petah Tikva
- Malaysia (2):
  - University Malaya Medical Centre, Lembah Pantai, Kuala Lumpur
  - Hospital Putrajaya, Putrajaya
- Consultorio de Endocrinología y Pediatría, Puebla City, Mexico
- Portugal (7):
  - Hospital Da Luz S.A., Lisbon
  - Hospital da Luz, Lisbon
  - Centro Hospitalar Lisboa Norte, Lisbon
  - Unidade Local De Saude De Santa Maria E.P.E., Lisbon
  - Unidade Local de Saúde de Santo António, E.P.E, Porto
  - CUF-Porto, Porto
  - Hospital CUF Porto S.A., Porto
- Russia (4):
  - FSBI 'I.I. Dedov National Medical Research Center of Endocrinology' of the MH of Russia, Moscow
  - NSMU paediatric clinic, Novosibirsk
  - Samara Regional Children Clinical Hospital n.a. N.N. Ivanova, Samara
  - Siberian State Medical University, Tomsk
- Switzerland (2):
  - Kantonsspital Olten, Olten
  - Kinderspital Endokrinologie, Zürich, Zurich

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Result] Fox CK, Barrientos-Perez M, Bomberg EM, Dcruz J, Gies I, Harder-Lauridsen NM, Jalaludin MY, Sahu K, Weimers P, Zueger T, Arslanian S; SCALE Kids Trial Group. Liraglutide for Children 6 to <12 Years of Age with Obesity - A Randomized Trial. N Engl J Med. 2025 Feb 6;392(6):555-565. doi: 10.1056/NEJMoa2407379. Epub 2024 Sep 10. PMID 39258838